CLINICAL TRIAL: NCT02821988
Title: Antenatal Testing in Obese Woman, is it Really Necessary?
Acronym: ATOWS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tennessee (Other)
Collaborators: Regional One Health (Other)
Responsible Party: Principal Investigator, Laura Grese, MD, University of Tennessee
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-04574-XP
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Obesity in Pregnancy
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Cardiotocography; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nonstress test (Experimental): Subjects will undergo weekly nonstress tests beginning at 32 weeks until delivery in addition to monitoring fetal kick counts.
  A nonstress test is a test in which an external fetal monitor is placed on the mother to defect the fetal heart rate for 20 to 40 minutes. A test is considered reactive if there are more than 2 accelerations in fetal heart rate defined as an increase of at least 15 beats per minute lasting at least 15 seconds in a 20 minute period.
  Interventions: Device: External fetal monitor for Nonstress test
- Biophysical profile (Experimental): Subjects will undergo weekly biophysical profile testing beginning at 32 weeks until delivery in addition to monitoring fetal kick counts. A Biophysical profile is a test using real time ultrasonography to determine the presence of absence of certain components of fetal well being. There components include: an episode of fetal breathing lasting at least 30 seconds, 3 or more discrete body movements, 1 or more episodes of extension of a fetal extremity with return to flexion, and determination of amniotic fluid volume to detect a maximum vertical pocket of >2cm. The duration of this test is no more than 30 minutes.
  Interventions: Device: Ultrasonography for Biophysical profile
- Kick counts only (No Intervention): Subjects will monitor fetal kick counts only.

INTERVENTIONS:
Device: External fetal monitor for Nonstress test
  Arms: Nonstress test
Device: Ultrasonography for Biophysical profile
  Arms: Biophysical profile

SUMMARY:
It is well established that obese women are at an increased risk of stillbirth compared to non obese women. This has led many physicians to begin antenatal testing in obese women in the third trimester through either nonstress tests or biophysical profiles. However, there is little evidence that antenatal testing improves fetal outcomes in obese women. The aim of this study is to determine if antenatal testing improves outcomes in obese women and to determine the optimal mode of testing (either nonstress tests or biophysical profiles).

DETAILED DESCRIPTION:
1. Purpose: To determine if antenatal testing improves outcomes in obese pregnant women
2. Rationale: It has been well established that obese pregnant women are at increase risk of stillbirth compared to matched non obese controls. This relative risk is increased not only with increasing gestational age in obese women but with increasing severity of obesity. The increased risk of stillbirth has led some obstetricians to begin antenatal testing in obese women; however, there is little evidence that antenatal fetal surveillance improves outcomes.
3. Study/Project Population: Pregnant women before 32 weeks of gestation with an initial BMI >30kg/m2
4. Research Design: Randomized Controlled Trial
5. Study/Project Procedures: Patients will be randomized to one of three groups: daily kick counts only, nonstress test, amniotic fluid index, and daily kick counts, and biophysical profile and daily kick counts. These patients will be randomly assigned a group in a 1:1:1 ratio using a random number generator available online. Patients assigned to the daily kick counts only group will be called weekly to ensure they are doing daily kick counts. If they are noncompliant, they will be removed from the study and will undergo nonstress tests if they meet the initial BMI criteria as is the standard practice at our institution.
6. Outcomes Measured: Stillbirth, induction of labor, mode of delivery, neonatal intensive care unit admission, AGPARs <7 at 5 minutes of life

ELIGIBILITY:
Inclusion Criteria:

less then 32 weeks gestation BMI > 30kg/m2 English speaking

Exclusion Criteria:

age < 18 age >45 medical comorbidity which requires antenatal testing other than obesity unwilling to consent Non-English speaking not pregnant Gestational age >32 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Stillbirth | until delivery, up to 41 weeks
  demise of infant prior to delivery as verified by ultrasonography
Mode of delivery | at delivery, up to 41 weeks
  whether the subject undergoes a vaginal delivery, cesarean delivery, or operative delivery will be recorded

SECONDARY OUTCOMES:
Neonatal intensive care unit admission admission | at delivery, up to 41 weeks
Apgar score of less than 7 at 5 minutes | at delivery, up to 41 weeks